CLINICAL TRIAL: NCT00844402
Title: Safety and Efficacy of Long-Term Treatment With Atorvastatin in Patients With Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Prof. Dr. Michael Trauner, Medical University of Graz, Department of Internal Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT_PBC-2
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Primary Biliary Cirrhosis; Hypercholesterolemia
Keywords: Cholestasis; Atherosclerosis; Statins; Vascular function
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Hypercholesterolemia; Cholestasis; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atorvastatin (Experimental): Atorvastatin 10 mg per day for 48 weeks
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — oral, 10 mg, daily, 48 weeks
  Other Names: Sortis10 mg, 1-21927, C10AA05

SUMMARY:
Primary biliary cirrhosis (PBC) is frequently associated with hypercholesterolemia and possibly with an increased cardiovascular morbidity and mortality. Statins lower serum cholesterol levels and may thus improve the cardiovascular risk in PBC patients. The aim of our study therefore was to prospectively examine the efficacy of low-dose atorvastatin on indicators of cardiovascular risk such as dyslipidemia and vascular function as well as safety in patients with PBC.

DETAILED DESCRIPTION:
Primary biliary cirrhosis (PBC) is often associated with abnormalities in serum lipids. Hypercholesterolemia is an established risk factor for cardiovascular morbidity and mortality. Since many PBC patients have a very slow progression of their underlying liver disease cardiovascular risk factors may become more relevant as prognostic facors. Whether statins lower serum cholesterol levels and reduce the cardiovascular risk in PBC patients remains to be determined. Statins are generally well tolerated and are not associated with an increased risk of hepatotoxicity in patients with nonalcoholic fatty liver disease (NAFLD). However only limited data on safety on statins in chronic cholestatic liver diseases are available. In a recent pilot study at the Medical University of Graz atorvastatin did not statistically increase liver enzymes in PBC patients. However, data on long-term treatment with atorvastatin in these patients are not yet available. Moreover, long-term treatment with statins may have potential beneficial immunomodulatory effects on the disease course of PBC in analogy to other immune-mediated disorders such as rheumatoid arthritis and multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* LDL-cholesterol > 130 mg/dl
* Primary biliary cirrhosis (AMA positive or biopsy proven)
* Male or female gender
* Age 18-70 years
* Normal kidney function

Exclusion Criteria:

* Primary biliary cirrhosis Stage III-IV (Ludwig Score)
* Liver cirrhosis
* Decompensated liver disease ( > Child-Pugh class B, ascites, esophageal varices)
* ALT or AST > 2x ULN
* Pregnancy or breastfeeding
* Premenopausal women without certain contraception
* Known hypersensitivity to HMG-CoA reductase inhibitors
* Current treatment with lipid-lowering agents other than atorvastatin; immunosuppressants, macrolides

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Low-density lipoprotein cholesterol (LDL-C) | week 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60

SECONDARY OUTCOMES:
Intima-media thickness of the common carotid artery (IMT), vascular wall stiffness (stiffness index SI), flow-mediated dilation of the brachial artery (FMD) | week 0, 48
Total cholesterol, triglycerides, VLDL-C, HDL-C, lipid profile, hs-CRP, AP, GGT, bilirubin, bile acids, immunoglobins | week 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60
AST, ALT, CK, PZ, AT, albumin, creatinine, blood cell count | week 0, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 60

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, M.D., Principal Investigator — Medical University of Graz, Department of Internal Medicine
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Derived] Stojakovic T, Claudel T, Putz-Bankuti C, Fauler G, Scharnagl H, Wagner M, Sourij H, Stauber RE, Winkler K, Marz W, Wascher TC, Trauner M. Low-dose atorvastatin improves dyslipidemia and vascular function in patients with primary biliary cirrhosis after one year of treatment. Atherosclerosis. 2010 Mar;209(1):178-83. doi: 10.1016/j.atherosclerosis.2009.08.052. Epub 2009 Sep 6. PMID 19782361